CLINICAL TRIAL: NCT06447402
Title: A Randomized Controlled Trial to Compare Nebulized Amphotericin B and Nebulized Normal Saline as Maintenance in Increasing Time to Relapse in Patients With Chronic Pulmonary Aspergillosis Treated With 12 Months of Oral Itraconazole
Brief Title: A Trial to Compare Nebulized Amphotericin B and Nebulized Normal Saline as Maintenance in Patients With Chronic Pulmonary Aspergillosis
Acronym: NAB-CPA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Inderpaul singh, Associate Professor, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SPL-577
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-06-10 (Actual); Status verified 2024-06

CONDITIONS: Chronic Pulmonary Aspergillosis; CPA; Aspergilloma
Keywords: CCPA; CFPA; CPA; Post TB lung abnormality; PTLD
MeSH Terms: interventions — Saline Solution; amphotericin B, deoxycholate drug combination

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Outcome assessor will be blinded to patient allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Saline arm (Placebo Comparator): 5 ml normal saline will be given as nebulization
  Interventions: Drug: Normal saline
- NAB arm (Experimental): Amphotericin B dexoycholate will be nebulised twice daily
  Interventions: Drug: Amphotericin B deoxycholate

INTERVENTIONS:
Drug: Normal saline — 5 mL of normal saline will be nebulised in the control arm
  Arms: Saline arm
Drug: Amphotericin B deoxycholate — 2 mL of the above reconstituted amphotericin B solution will be obtained in a sterile syringe and transferred into the drug chamber of a nebulizer. Three mL of distilled water will be added to 2 mL of the reconstituted amphotericin B (5 mL liquid in the chamber ensures complete and easy nebulization of all the contents)
  Arms: NAB arm

SUMMARY:
The treatment of CPA is with oral itraconazole for 6-12 months. Oral itraconazole results in better clinical outcomes in CPA compared to supportive care. A recent study comparing 6 months with 12 months of oral itraconazole for longer duration treatment found longer duration reduced CPA relapse and improved clinical outcomes. However, longer duration of itraconazole could cause emergence of drug resistant Aspergillus fumigatus and therapy related adverse event. A recent study found nebulized amphotericin B non-inferior to oral itraconazole for treating CPA as primary therapy. However, the study was small and included patients with simple aspergilloma and used nebulized amphotericin B for 7 days.To be effective, an inhaled drug should be delivered in sufficient quantity to achieve therapeutic levels.The minimum inhibitory concentration of amphotericin B for A.fumigatus is 0.5 mg/L. In one study, nebulization of 30 mg of amphotericin B deoxycholate achieved a mean concentration of 0.68 mg/L in the bronchoalveolar lavage fluid. Notably, the serum levels of amphotericin B after nebulization are 20 times less than after systemic administration and is safer. Further, there is a dose-response relation with nebulized amphotericin B, the higher the dose used for nebulization, the higher are the levels achieved in the lung tissue. Nebulized amphotericin B has been used in lung transplant recipients to prevent invasive aspergillosis. Also, two recent studies have demonstrated that use of nebulized amphotericin B as maintenance therapy led to a reduction in ABPA relapse rates and prolonged time to exacerbation. We believe that inhaled amphotericin B as a maintenance therapy could reduce CPA relapse and prolong time to relapse. In this study, we plan to evaluate nebulized amphotericin B as a maintenance therapy in clinically stable CPA patients treated with 12 months of oral antifungal therapy

DETAILED DESCRIPTION:
Aspergillus is a ubiquitous fungus that causes a spectrum of human lung diseases depending on the host immunity and the immune response. In those with overt immunodeficiency, Aspergillus spp. causes invasive pulmonary aspergillosis. In immunocompetent individuals with structurally damaged lungs Aspergillus spp. causes chronic pulmonary aspergillosis. On the other hand, allergic bronchopulmonary aspergillosis (ABPA) complicated the disease course of asthmatics and cystic fibrosis due to a hyperimmune response mounted by the host against the fungi colonizing the airways.

Chronic pulmonary aspergillosis (CPA) has significant global burden, yet under-reported aspergillus related chronic lung disease. CPA is a chronic progressive lung disease that has a five-year mortality of over 50%. CPA has a significant global burden with more than a million individuals are affected with CPA globally. In India alone, more than 100,000 individuals are affected with CPA annually. CPA occurs primarily in patients with pre-existing structural lung disease, including post-pulmonary tuberculosis lung disease (PTBLD), chronic obstructive pulmonary disease (COPD), and others. In our experience, PTBLD is the most common risk factor for CPA.(3-5) While the treatment of pulmonary TB is highly effective, almost 25-30% of the cases are left with sequelae of the disease including cavities, parenchymal fibrosis, and others. Patients with sequelae are not only at higher risk of recurrence of TB but are also prone to colonization with Aspergillus fumigatus. It has been estimated that CPA develops in approximately 20-25% of treated pulmonary tuberculosis with residual cavity. Unfortunately, the recognition of CPA is poor amongst physicians and even pulmonary physicians. Patients with recurrent cough, hemoptysis, fever or weight loss and a negative sputum examination for AFB or Xpert MTB/Rif are labelled as smear negative pulmonary tuberculosis. In fact, almost 50% of the patients with CPA are misdiagnosed as pulmonary TB and receive empiric anti-TB therapy because of the similarities in presentation of the two disorders. Untreated CPA is fatal with a five-year mortality of 30-80%.This has clinical implications as these patients with CPA would benefit from antifungal agents. While the actual burden of CPA among treated TB patients is not known, a mathematical model estimated that approximately 0.14 million cases are affected annually. Further, it was shown that if the mortality of CPA is estimated as 15% annually, the 5-year burden of CPA is about 290,147 cases with a 5-year prevalence rate of 24 per 100,000.

The diagnosis of CPA is based on the constellation of clinical symptoms (low-grade fever, weight loss, anorexia, malaise, cough with expectoration, recurrent hemoptysis, fatigue, chest pain, and dyspnea, for at least three months), persistent or progressive radiological features (one or more cavities with or without fungal ball, fibrosis, pericavitary infiltrates, consolidation, nodules and pleural thickening) and the presence of either direct (positive sputum or bronchoalveolar lavage fluid [BALF] culture) or indirect (elevated serum or BALF galactomannan index or Aspergillus fumigatus-specific precipitins [or IgG] antibodies in serum) evidence of Aspergillus infection. Of the available diagnostic modalities, serology is the most reliable component of the CPA diagnostic pathway. Currently, the estimation of A.fumigatus-specific IgG by enzyme immunoassay (Phadia, Immulite and others) is considered the most sensitive test in the diagnosis of CPA. In a recent study, using a cut-off of 27 mgA/L, the sensitivity of A.fumigatus-specific IgG in the diagnosis of CPA was about 91.3%.The prevalence of CPA in India in subjects not known. Our group has estimated the burden of CPA following pulmonary TB using a mathematical modelling.

The treatment of CPA is with oral itraconazole for 6-12 months. Oral itraconazole results in better clinical outcomes in CPA compared to supportive care. A recent study comparing 6 months with 12 months of oral itraconazole for longer duration treatment found longer duration reduced CPA relapse and improved clinical outcomes. However, longer duration of itraconazole could cause emergence of drug resistant Aspergillus fumigatus and therapy related adverse event. A recent study found nebulized amphotericin B non-inferior to oral itraconazole for treating CPA as primary therapy. However, the study was small and included patients with simple aspergilloma and used nebulized amphotericin B for 7 days.To be effective, an inhaled drug should be delivered in sufficient quantity to achieve therapeutic levels. The minimum inhibitory concentration of amphotericin B for A.fumigatus is 0.5 mg/L. In one study, nebulization of 30 mg of amphotericin B deoxycholate achieved a mean concentration of 0.68 mg/L in the bronchoalveolar lavage fluid. Notably, the serum levels of amphotericin B after nebulization are 20 times less than after systemic administration and is safer. Further, there is a dose-response relation with nebulized amphotericin B, the higher the dose used for nebulization, the higher are the levels achieved in the lung tissue. Nebulized amphotericin B has been used in lung transplant recipients to prevent invasive aspergillosis. Also, two recent studies have demonstrated that use of nebulized amphotericin B as maintenance therapy led to a reduction in ABPA relapse rates and prolonged time to exacerbation. We believe that inhaled amphotericin B as a maintenance therapy could reduce CPA relapse and prolong time to relapse. In this study, we plan to evaluate nebulized amphotericin B as a maintenance therapy in clinically stable CPA patients treated with 12 months of oral antifungal therapy.

AIMS To compare the clinical outcomes of nebulized amphotericin B deoxycholate versus nebulized normal saline as maintenance therapy in CPA subjects treated with 12 months of antifungal therapy

ELIGIBILITY:
Inclusion Criteria:

* consecutive subjects with CPA who have received 12 months therapy with oral itraconazole

Exclusion Criteria:

(i) failure to provide informed consent; (ii) patients on immunosuppressive drugs, intake of >10 mg prednisolone (or equivalent) for at least 3 weeks in last 3 months, or a diagnosis of human immunodeficiency virus syndrome, ; (iii) subjects with active pulmonary infection due to mycobacterium tuberculosis or mycobacteria other than tuberculosis (MOTT); (iv) subjects with others forms of pulmonary aspergillosis (subacute and acute invasive aspergillosis); (v) pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2026-06-03 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to first exacerbation | 12 months after randomization
  Time to exacerbation of CPA after stopping itraconazole

SECONDARY OUTCOMES:
frequency of relapses at 12-months after randomization | 12 months after randomization
  number of CPA relapsed during follow up
Treatment emergent adverse events | 12 months after randomization
  Number of therapy related adverse reactions in each arm

CONTACTS AND LOCATIONS:
Locations (1):
- Chest clinic, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Undecided
We will share on a reasonable request to the PI